CLINICAL TRIAL: NCT06415773
Title: A Phase 3, Multicenter, Randomized, Double-Blind, Active-Controlled (Dapagliflozin), Parallel Group Efficacy and Safety Study of HTD1801 in Patients With Type 2 Diabetes Mellitus Inadequately Controlled With Metformin Alone
Brief Title: Effects of Berberine Ursodeoxycholate (HTD1801) Versus Dapagliflozin in Patients With Type 2 Diabetes Inadequately Controlled With Metformin
Acronym: HARMONY
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: HighTide Biopharma Pty Ltd (Industry)
Collaborators: Shenzhen HighTide Biopharmaceutical Ltd. (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: HTD1801.PCT109
Record Dates: First submitted 2024-05-10; First posted 2024-05-16 (Actual); Last update posted 2025-12-31 (Actual); Status verified 2025-12

CONDITIONS: T2DM (Type 2 Diabetes Mellitus)
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — dapagliflozin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- HTD1801 (Experimental): Administered orally twice daily (BID)
  Interventions: Drug: HTD1801
- Dapagliflozin (Active Comparator): Administered orally once daily (QD)
  Interventions: Drug: Dapagliflozin

INTERVENTIONS:
Drug: HTD1801 — HTD1801 1000 mg BID administered orally BID as four capsules
  Other Names: Berberine Ursodeoxycholate
  Arms: HTD1801
Drug: Dapagliflozin — Dapagliflozin 10 mg tablet administered orally QD
  Arms: Dapagliflozin

SUMMARY:
The goal of this clinical study is to evaluate the efficacy and safety of berberine ursodeoxycholate (HTD1801) compared to dapagliflozin in patients with type 2 diabetes inadequately controlled with metformin alone.

DETAILED DESCRIPTION:
This Phase 3 randomized, double-blind, active-controlled, parallel-group study will evaluate the efficacy and safety of HTD1801 compared to dapagliflozin after 24 weeks of treatment. All patients will remain on a stable dose of metformin throughout the study.

To ensure stabilization of glycemic control, eligible patients will first participate in a 4-week single-blind run-in period where investigators will provide guidance on lifestyle modification, concomitant medications, and procedures for self-monitoring of blood glucose. Following this period, patient eligibility will be reassessed. Eligible patients will then be randomized 1:1 to receive HTD1801 1000 mg BID or dapagliflozin 10 mg QD.

ELIGIBILITY:
Inclusion Criteria:

* Have been diagnosed with type 2 diabetes
* Have received a stable dose of metformin monotherapy for at least 8 weeks prior to screening
* If used any glucose-lowering drugs other than metformin within the 8 weeks prior to screening such use was ≤7 days and was discontinued at least 4 weeks prior to screening
* Have HbA1c ≥7.5% to ≤11.0% (screening) and HbA1c ≥7.0% to ≤10.5% (pre-randomization)
* Have fasting plasma glucose ≤13.9 mmol/L (screening and pre-randomization)
* Have a body mass index ≥19.0 kg/m^2 and ≤35.0 kg/m^2

Exclusion Criteria:

* Have type 1 diabetes
* Have had any acute diabetic complications within 12 months prior to screening
* Have had any Grade 3 hypoglycemic event within 12 months prior to screening
* Have had proliferative retinopathy or macular degeneration, severe diabetic neuropathy, or diabetic foot
* Have been taking any weight loss medication or dietary supplement, have participated in a weight loss program, or have adhered to a special diet within 12 weeks prior to screening
* Have used insulin or an insulin analogue for more than 14 days within 12 months prior to screening
* Have used any hypoglycemic drug other than metformin during the 4-week run-in period prior to randomization
* Have had weight gain or loss ≥5% during the 4-week run-in period prior to randomization
* Have a history of refractory or recurrent urinary tract infections or genital infections

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 367 (Actual)
Dates: Start 2024-06-04 (Actual); Primary Completion 2025-06-13 (Actual); Study Completion 2025-07-25 (Actual)

PRIMARY OUTCOMES:
Primary Endpoint: Mean change in HbA1c | 24 Weeks
  Mean change in HbA1c from baseline to Week 24

SECONDARY OUTCOMES:
Mean Change in Fasting Plasma Glucose | 24 Weeks
  Mean change in fasting plasma glucose from baseline to Week 24
Mean Change in 2-Hour Postprandial Glucose | 24 Weeks
  Mean change in 2-hour postprandial glucose from baseline to Week 24
Proportion of Patients Achieving HbA1c <7.0% | 24 Weeks
  Proportion of patients achieving HbA1c <7.0% after 24 weeks of treatment
Proportion of Patients Achieving HbA1c <6.5% | 24 Weeks
  Proportion of patients achieving HbA1c <6.5% after 24 weeks of treatment
Mean Change in Insulin Sensitivity (HOMA-IR) | 24 Weeks
  Mean change in homeostatic model assessment for insulin resistance (HOMA-IR) from baseline to Week 24
Mean Change in Low-Density Lipoprotein Cholesterol (LDL-C) | 24 Weeks
  Mean change in LDL-C from baseline to Week 24

CONTACTS AND LOCATIONS:
Overall Officials: Kui Liu, MD, Study Director — Shenzhen HighTide Biopharmaceutical Ltd.
Locations (53):
- China (53):
  - Beijing Pinggu Hospital, Beijing
  - Peking University People's Hospital, Beijing
  - Binzhou Medical University Hospital, Binzhou
  - Jilin Province FAW General Hospital, Changchun
  - The Second Hospital of Jilin University, Changchun
  - The First People's Hospital of Changde City, Changde
  - The First Hospital of Changsha City, Changsha
  - The Fourth Hospital of Changsha, Changsha
  - The Second Xiangya Hospital of Central South University, Changsha
  - The Third Xiangya Hospital of Central South University, Changsha
  - Bishan Hospital of Chongqing, Chongqing
  - People's Hospital of Deyang City, Deyang
  - Handan First Hospital, Handan
  - The Fourth Hospital of Harbin Medical University, Harbin
  - The Second People's Hospital of Huai'an, Huai'an
  - Huanggang Central Hospital, Huanggang
  - Huangshi Central Hospital, Huangshi
  - Huizhou Municipal Central Hospital, Huizhou
  - Jincheng General Hospital, Jincheng
  - Hebei Petro China Central Hospital, Langfang
  - The Second People's Hospital of Lianyungang, Lianyungang
  - Liaocheng People's Hospital, Liaocheng
  - Luoyang Third People's Hospital, Luoyang
  - The First Affiliated Hospital of Henan University of Science & Technology (Jinghua), Luoyang
  - The First Affiliated Hospital of Henan University of Science & Technology (Kaiyuan), Luoyang
  - The First Affiliated Hospital of Nanchang University, Nanchang
  - The Second Affiliated Hospital of Nanchang University, Nanchang
  - Nanjing Drum Tower Hospital - The Affiliated Hospital of Nanjing University Medical School, Nanjing
  - The Second Affiliated Hospital of Nanjing Medical University, Nanjing
  - Affiliated Hospital of Nantong University, Nantong
  - The First Affiliated Hospital of Nanyang Medical College, Nanyang
  - Panjin Liaohe Oilfield GEM Flower Hospital, Panjin
  - Pingxiang People's Hospital, Pingxiang
  - The First Hospital of Qiqihar, Qiqihar
  - Sanmenxia Central Hospital, Sanmenxia
  - Huadong Hospital Affiliated to Fudan University, Shanghai
  - Shanghai Sixth People's Hospital, Shanghai
  - Shengjing Hospital of China Medical University, Shenyang
  - The People's Hospital of Liaoning Province, Shenyang
  - Wuhan Third Hospital, Wuhan
  - The First Affiliated Hospital of Xi'an Jiaotong University, Xi'an
  - The Second Affiliated Hospital of Xi'an Jiaotong University, Xi'an
  - The Central Hospital of Xiangtan, Xiangtan
  - The First People's Hospital of Xiangtan City, Xiangtan
  - Xianyang Hospital of Yan'an University, Xianyang
  - Xuzhou Cancer Hospital, Xuzhou
  - The Second People's Hospital of Yibin, Yibin
  - Yiyang Central Hospital, Yiyang
  - Yueyang People's Hospital, Yueyang
  - Shandong Guoxinyiyang Group Zaozhuang Central Hospital, Zaozhuang
  - The Second Affiliated Hospital of Zhengzhou University, Zhengzhou
  - Affiliated Hospital of Jiangsu University, Zhenjiang
  - Zhumadian Central Hospital, Zhumadian

IPD SHARING:
Plan to Share IPD: No